CLINICAL TRIAL: NCT01553084
Title: A Comparative Effectiveness & Long Term Health Study in Wisconsin Smokers
Acronym: NHLBI-RO1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01HL109031-01 (NIH); 1R01HL109031-01 (NIH); 2011-0756 (Other: UW, Madison)
Record Dates: First submitted 2011-11-09; First posted 2012-03-13 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation; Smoking; Nicotine Dependence
Keywords: Smoking Cessation; Smoking; Nicotine
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Disorder | interventions — Varenicline; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Effectiveness of Nicotine patch only (Experimental)
  Interventions: Drug: Nicotine Patch
- Effectiveness of Combination NRT (Experimental)
  Interventions: Drug: Nicotine lozenge; Drug: Nicotine Patch
- Effectiveness of Varenicline [Chantix] (Experimental)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Participants will receive 12 weeks of pharmacotherapy during the post-quit period plus an additional 7 day pre-quit run-in. Participants will be asked to take a 0.5 mg pill once a day for the first 3 days and then increase to a 0.5 mg pill twice a day (8 hours apart) for 4 days. On the 8th day, their target quit date, they will increase to their target maintenance dose of a 1 mg pill twice daily. If participants report significant adverse events such as nausea, a dose reduction to two 0.5 mg doses per day will be advised.
  Arms: Effectiveness of Varenicline [Chantix]
Drug: Nicotine lozenge — Participants will receive 12 weeks NRT. Participants will be given 2 mg or 4 mg lozenges based on morning smoking latency, and will be given package insert use instructions. Medication use will start on the morning of their assigned quit day. They will be urged to use at least 5 pieces/day, unless this amount produces adverse effects.
  Arms: Effectiveness of Combination NRT
Drug: Nicotine Patch — Participants will receive 12 weeks NRT. Patch dosing will be 8 weeks of 21 mg, then 2 weeks of 14 mg, then 2 weeks of 7 mg (those smoking 5-10 cigs/day will receive reduced patch dosing). Medication use will start on the morning of their assigned quit day. They will be urged to use 1 patch/day, unless it produces adverse effects.
  Arms: Effectiveness of Combination NRT; Effectiveness of Nicotine patch only

SUMMARY:
The overall purpose of this research is two-fold. First, the two smoking cessation medication treatments with the strongest evidence of effectiveness have never been directly compared. This research will determine how these two treatments compare in effectiveness in a head-to-head trial, and which types of smokers benefit most from each. Second, much of the data on smoking and health come from studies from many years ago. Today's smokers differ from earlier smokers in many ways that could influence the impact of smoking on health (e.g., weight, sex, diet, socio-economic status); the proposed work will determine how smoking cessation affects cardiovascular and pulmonary health in today's smokers.

DETAILED DESCRIPTION:
The proposed study will recruit and treat a large sample of contemporary smokers and former smokers at an age of increasing health risk, to achieve the following over-arching aims that are important to the NHLBI mission:

* Specific Aim 1: Produce important new data on how to treat smoking optimally by conducting an open label comparative effectiveness trial (CET) that for the first time directly contrasts the two smoking cessation pharmacotherapies with the strongest extant evidence of efficacy: combination NRT and varenicline.
* Specific Aim 2: Determine the impact of smoking cessation on biomarkers and health risk factors, especially those relevant to CVD, in today's smokers, which will elucidate the mechanisms via which cessation benefits health.
* Specific Aim 3: Identify which individuals are at greatest risk for exacerbation of biomarkers or risk factor status due to continued smoking, and who will benefit most from cessation. This will help identify individuals who are most in need of cessation intervention. While all smokers need to quit, this evidence could ultimately be used to help focus treatment and motivate smokers and clinicians to intervene more intensively with patients at greatest risk.

Two secondary aims are to use the results of Primary Aim 1 to develop a treatment assignment algorithm for the optimal treatment of today's smokers and to use the results from Primary Aim 2 to determine the relation of health biomarkers to clinically meaningful disease outcomes such as CVD events.

We will re-recruit as many smoking and non smoking participants from our past longitudinal cohort study("Wisconsin Smokers' Health study"; NCT01122238) in 2004. We will then recruit additional smokers to participate in the comparative effectiveness trial and join the longitudinal cohort..

All participants who enroll will complete questionnaires about their demographics, smoking history, withdrawal symptoms, affect, alcohol use, stressors, medication usage and diet. They will also complete a structured clinical interview to assess mental health. They will provide blood samples for testing of various markers of cardiovascular disease and risk as well as for genetics testing. They will all have carotid ultrasounds, pulmonary function tests, arterial tonometry assessments, and 12-lead ECGs. Participants in Madison will also have a treadmill stress test. Participants will wear a pedometer for 1 week and record the daily number of steps. Participants will provide permission for staff to review their medical charts to assess smoking-relevant diagnoses and treatment. These assessments will occur at baseline and again 3 years later. A smaller subset of these assessments will also be conducted 1 year after enrollment. Participants will also complete brief phone assessments at 6-month intervals up to the 3-year visit.

Interested and eligible smoking participants from the original cohort study and all newly recruited participants will enroll in a new smoking cessation intervention study. Participants in the cessation treatment study will be randomly assigned to receive the nicotine patch, nicotine patch + nicotine lozenge or varenicline. If the participant from the original cohort study is not eligible to use all study medications but is otherwise eligible for cessation treatment, s/he will be assigned to a non-randomized treatment arm and will receive nicotine patch (if appropriate). All cessation participants will receive 6 individual counseling sessions.

ELIGIBILITY:
We are only recruiting by invitation only (to members of our past cohort). We will open up enrollment to the public in the Madison, WI and Milwaukee WI areas at the end of 2012.

Inclusion Criteria:

a. To be eligible for the Comparative effectiveness trial, participants must:

* smoke 5 or more cigarettes per day,
* desire to quit smoking but not be currently engaged in cessation treatment,
* be medically eligible to use either combination NRT or varenicline,
* have reliable phone access,
* if female, must not be pregnant and must be willing to use an acceptable birth control method.

Exclusion Criteria:

1. There are no exclusion criteria for participating in the main health outcomes study, other than being unwilling to complete study assessments.
2. All smoking participants from new and original cohorts will be excluded from the cessation trial for the following reasons:

   * end-stage renal disease with hemodialysis;
   * prior suicide attempts within the last 5 years or current suicidal ideation;
   * diagnosis of and/or treatment for schizophrenia;
   * other psychotic disorders or bipolar disorder within the last 10 years;
   * current PHQ-9 score indicative of moderately severe depression;
   * severe untreated hypertension >200/100 mmHg;
   * currently taking Wellbutrin, Zyban or bupropion;
   * hospitalized for a stroke, heart attack, congestive heart failure or diabetes within the last year;
   * used pipe tobacco, cigars, snuff or chew more than twice in the past week.

It should be noted that if any incidental findings appear in any of the cardiology tests (e.g., ultrasound, tonometry, ECG, or exercise stress test; see forms in Supplemental Information section of application), the study cardiologist (Dr. Stein or his designee) will be assign the participant to the non-randomized treatment arm and they will be given the nicotine patch and the same counseling intervention as CET participants. They will not be included in the CET analyses. This will be done to properly address the cardiovascular risk warning from the FDA regarding varenicline (Chantix).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1086 (Actual)
Dates: Start 2012-05; Primary Completion 2015-11 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Fiore, MD, MPH, Principal Investigator — University of Wisconsin, Madison; James H Stein, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin
  - University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Milwaukee, Wisconsin

REFERENCES:
- [Result] Baker TB, Piper ME, Stein JH, Smith SS, Bolt DM, Fraser DL, Fiore MC. Effects of Nicotine Patch vs Varenicline vs Combination Nicotine Replacement Therapy on Smoking Cessation at 26 Weeks: A Randomized Clinical Trial. JAMA. 2016 Jan 26;315(4):371-9. doi: 10.1001/jama.2015.19284. PMID 26813210
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Karim R, Xu W, Kono N, Sriprasert I, Li Y, Yan M, Stanczyk FZ, Shoupe D, Mack WJ, Hodis HN. Effect of menopausal hormone therapy on arterial wall echomorphology: Results from the Early versus Late Intervention Trial with Estradiol (ELITE). Maturitas. 2022 Aug;162:15-22. doi: 10.1016/j.maturitas.2022.02.007. Epub 2022 Mar 17. PMID 35474254
- [Derived] Kaye JT, Johnson AL, Baker TB, Piper ME, Cook JW. Searching for Personalized Medicine for Binge Drinking Smokers: Smoking Cessation Using Varenicline, Nicotine Patch, or Combination Nicotine Replacement Therapy. J Stud Alcohol Drugs. 2020 Jul;81(4):426-435. doi: 10.15288/jsad.2020.81.426. PMID 32800078
- [Derived] Mitchell C, Piper ME, Smith SS, Korcarz CE, Fiore MC, Baker TB, Stein JH. Changes in carotid artery structure with smoking cessation. Vasc Med. 2019 Dec;24(6):493-500. doi: 10.1177/1358863X19867762. Epub 2019 Aug 17. PMID 31422759
- [Derived] Schlam TR, Baker TB, Smith SS, Cook JW, Piper ME. Anxiety Sensitivity and Distress Tolerance in Smokers: Relations With Tobacco Dependence, Withdrawal, and Quitting Successdagger. Nicotine Tob Res. 2020 Jan 27;22(1):58-65. doi: 10.1093/ntr/ntz070. PMID 31056710
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix]
Started | 241 | 421 | 424
Completed | 226 | 408 | 389
Not Completed | 15 | 13 | 35
Not completed — Withdrawal by Subject | 15 | 13 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix] | Total
Number analyzed (Participants) | 241 | 421 | 424 | 1086
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (10.9) | 47.1 (11.7) | 48.5 (11.8) | 48.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 219 | 222 | 566
  Male | 116 | 202 | 202 | 520
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 1 | 6
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 72 | 117 | 120 | 309
  White | 158 | 287 | 283 | 728
  More than one race | 6 | 5 | 11 | 22
  Unknown or Not Reported | 2 | 7 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 241 | 421 | 424 | 1086

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-confirmed 7-Day Point-Prevalence Abstinence at 26 Weeks
Description: Self-reported total abstinence from any tobacco use (even a single puff) for the seven days preceding the target follow-up day, confirmed with an exhaled carbon monoxide reading of <10 ppm..
Time Frame: Assessed 26 weeks after the target quit day.
Measure: Count of Participants; unit: Participants
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix]
Number analyzed (Participants) | 241 | 421 | 424
Participants | 63 | 124 | 108
Statistical Analysis 1: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Combination NRT; Combination NRT will be compared statististically versus Nicotine patch only (the reference or control group); Test type: Superiority; p = .3623, Regression, Logistic; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.8 to 1.7]
Statistical Analysis 2: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Varenicline [Chantix]; Varenicline will be compared statististically versus Nicotine patch only (the reference or control group); Test type: Superiority; p = .1947, Regression, Logistic; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.6 to 1.2]

2. Secondary Outcome: Number of Days to Relapse
Description: The number of days to relapse is defined as the number of days from the target quit day until the first of seven consecutive days of smoking.
Time Frame: Assessed from the target quit day through 26 weeks.
Population: Participants who did not relapse were censored in the survival analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix]
Number analyzed (Participants) | 241 | 421 | 424
Days | 29.3 (42.4) | 37.4 (46.5) | 31.7 (46.7)
Statistical Analysis 1: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Combination NRT; Test type: Superiority; p = .3613, Regression, Cox; Hazard Ratio (HR) = .915, 95% CI 2-sided [.756 to 1.107]
Statistical Analysis 2: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Varenicline [Chantix]; Test type: Superiority; p = .5503, Regression, Cox; Hazard Ratio (HR) = .943, 95% CI 2-sided [.779 to 1.142]

3. Secondary Outcome: Number of Participants With Initial Cessation in the First 7 Days Post-quit
Description: Defined as at least 1 day of abstinence during the first 7 days after the target quit day.
Time Frame: Assessed for the first seven days after the target quit date.
Measure: Count of Participants; unit: Participants
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix]
Number analyzed (Participants) | 241 | 421 | 424
Participants | 176 | 339 | 289
Statistical Analysis 1: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Combination NRT; Test type: Superiority; p = .03, Regression, Logistic; Odds Ratio (OR) = 1.5, 95% CI 2-sided [1.1 to 2.2]
Statistical Analysis 2: Comparison: Effectiveness of Nicotine Patch Only vs Effectiveness of Varenicline [Chantix]; Test type: Superiority; p = .19, Regression, Logistic; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.6 to 1.1]

4. Secondary Outcome: The Effects of Quitting Smoking vs. Continued Smoking on Change in Carotid Intima-media Thickness (CIMT).
Description: Change in carotid intima-media thickness (CIMT) from Baseline to Year 3 as a function of smoking status (abstinent versus smoking) at Year 3. Change is calculated as Baseline CIMT score minus Year 3 CIMT score. CIMT score is thickness of the carotid intima-media in millimeters (mm). Lower CIMT values indicate a better outcome.
Time Frame: Assessed at Baseline and Year 3
Population: Includes only participants who completed both Baseline and Year 3 CIMT measurements.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Groups:
- Abstinent at Year 3: Participants who are abstinent at Year 3 with biochemical confirmation.
- Smoking at Year 3: Participants who are smoking at Year 3.
Arm/Group | Abstinent at Year 3 | Smoking at Year 3
Number analyzed (Participants) | 190 | 522
millimeters (mm) | -0.0682 (0.0689) | -0.0620 (0.0755)
Statistical Analysis 1: Comparison: Abstinent at Year 3 vs Smoking at Year 3; Test type: Superiority; p = .3282, t-test, 2 sided; df=710; Mean Difference (Final Values) = -0.00612, Standard Error of Mean 0.00625

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12 weeks while participants were taking study medication.
Description: Study participants were asked: "Since your last contact with us, has there been any change in your medical condition or health?" at 1 week prior to the quit smoking visit (quit day), on the quit day, at week 1, week 4, week 8, and week 12. Participants also could self-initiate symptom reports during other visits or phone calls. Information on All-Cause Mortality was not collected.
Arm/Group | Effectiveness of Nicotine Patch Only | Effectiveness of Combination NRT | Effectiveness of Varenicline [Chantix]
All-Cause Mortality (participants affected / at risk) | 5/241 | 6/421 | 5/424
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/421 | 1/424
Other Adverse Events (participants affected / at risk) | 164/241 | 281/421 | 353/424
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Effectiveness of Nicotine Patch Only (N=241) | Effectiveness of Combination NRT (N=421) | Effectiveness of Varenicline [Chantix] (N=424)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Effectiveness of Nicotine Patch Only (N=241) | Effectiveness of Combination NRT (N=421) | Effectiveness of Varenicline [Chantix] (N=424)
Itching/hives (Immune system disorders) | 53 (53) | 74 (74) | 7 (7)
Vivid Dreams (Psychiatric disorders) | 40 (40) | 55 (55) | 98 (98)
Insomnia (Psychiatric disorders) | 35 (35) | 45 (45) | 94 (94)
Rash (Skin and subcutaneous tissue disorders) | 27 (27) | 48 (48) | 9 (9)
Nausea (Gastrointestinal disorders) | 20 (20) | 62 (62) | 121 (121)
Vomiting (Gastrointestinal disorders) | 6 (6) | 13 (13) | 22 (22)
Constipation (Gastrointestinal disorders) | 5 (5) | 13 (13) | 29 (29)
Dizziness (Nervous system disorders) | 18 (18) | 20 (20) | 27 (27)
Headache (Nervous system disorders) | 15 (15) | 28 (28) | 29 (29)
Sleepiness (General disorders) | 10 (10) | 26 (26) | 68 (68)
Indigestion (Gastrointestinal disorders) | 4 (4) | 42 (42) | 22 (22)
Mouth Problems (Product Issues) | 3 (3) | 33 (33) | 7 (7)
Hiccups (Gastrointestinal disorders) | 0 (0) | 26 (26) | 1 (1)
Heart Symptoms (Cardiac disorders) | 14 (14) | 13 (13) | 26 (26) — Chest tightness, angina (heart pain), shortness of breath.
Depression (Psychiatric disorders) | 10 (10) | 13 (13) | 25 (25) — Feeling depressed or hopeless.
Anxious (Psychiatric disorders) | 18 (18) | 26 (26) | 20 (20) — Feeling worried, nervous, scared or anxious.
Agitated/restless (Psychiatric disorders) | 15 (15) | 14 (14) | 35 (35) — Feeling agitated or restless.
Hostile/angry (Psychiatric disorders) | 7 (7) | 11 (11) | 23 (23) — Feeling hostile or angry towards others.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No